CLINICAL TRIAL: NCT02900924
Title: A Prospective, Multicentre Observational Study to Evaluate the BioMimics 3D Self-Expanding Stent System in the Treatment of Peripheral Arterial Disease: MIMICS-3D
Brief Title: Observational Study to Evaluate the BioMimics 3D Stent System: MIMICS-3D
Acronym: MIMICS-3D
Status: Completed | Type: Observational
Sponsor: Veryan Medical Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: MIMICS-3D
Record Dates: First submitted 2016-08-25; First posted 2016-09-15 (Estimated); Results first posted 2025-04-17 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-03

CONDITIONS: Peripheral Arterial Disease
Keywords: PAD; PVD; SFA stent
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: BioMimics 3D Stent

SUMMARY:
The MIMICS-3D study will evaluate safety, effectiveness and device performance within a real-world clinical population of patients undergoing femoropopliteal intervention.

DETAILED DESCRIPTION:
The MIMICS-3D study is a prospective, multicentre, observational study of the BioMimics 3D Stent System in patients undergoing endovascular intervention to relieve symptomatic peripheral arterial disease of the femoropopliteal artery. The study is designed to enable the collection, analysis and reporting of data from "real-world" use of the BioMimics 3D Stent System used in accordance with the Instructions for Use (IFU) associated with the product's CE Mark approval.

Data collection will include that relating to safety, effectiveness and device performance and the period of observation during which data will be collected will extend from the index procedure through 3 years (36 months), according to the standard follow-up practice of the enrolling institution.

ELIGIBILITY:
Inclusion Criteria:

* Patient is age ≥18 and ≤85 years at date of consent.
* Patient has provided written informed consent for participation in the study prior to index procedure.
* Patient has documented symptomatic peripheral arterial disease scheduled for treatment with the BioMimics 3D stent in accordance with the approved CE Mark indication and Instructions for Use (IFU)

Exclusion Criteria:

* Patients whose lesions cannot be crossed with a wire and/or balloon catheter and cannot be dilated sufficiently to allow passage of the delivery system.
* Patients with a history of intolerance or adverse reaction to antiplatelet and/or anticoagulation therapies, bleeding diathesis, severe hypertension or renal failure.
* Patients with known hypersensitivity to nickel-titanium.
* Patient has a comorbidity that in the Investigator's opinion would limit life expectancy to less than 12 months.
* Patient is pregnant or breastfeeding.
* Patient is unable or is unwilling to comply with site standard of care procedures and follow-up visit schedules for patients undergoing femoropopliteal intervention.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who receive treatment with Veryan's BioMimics 3D Stent System in accordance with the current approved CE Mark indication for use as stated in the Instructions for Use (IFU) will be consecutively enroled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 507 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2019-10 (Actual); Study Completion 2021-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Lichtenberg, MD, Principal Investigator — Klinikum Arnsberg
Locations (23):
- Belgium (5):
  - OLV Hospital, Aalst
  - ZNA Vascular Clinic/ZNA Stuivenburg Hospital, Antwerp
  - AZ Sint Blasius, Dendermonde
  - AZ Maria Middelares, Ghent
  - Regionaal Vaartcentrum , AZ Helig Hart Tienen, Tienen
- Germany (16):
  - Karolinen-Hospital, Arnsberg
  - Universitaets-Herzzentrum Freiburg-Bad Krozingen, Bad Krozingen
  - KEH Berlin, Berlin
  - Vivantes Klinikum Friedrichshain, Berlin
  - Krankenhaus Buchholz, Buchholz
  - Krankenhaus Dresden-Friedrichstadt, Städtisches Klinikum, Dresden
  - Universitätsklinikum Essen, Essen
  - CCB im Agaplesion Bethanien Krankenhaus, Frankfurt am Main
  - Asklepios Klinik Harburg, Hamburg
  - UKE (University Hospital Hamburg), Hamburg
  - Universitätsklinikum Leipzig AöR, Leipzig
  - Gefäßpraxis im Tal, Munich
  - Marienhospital Osnabrück GmbH, Osnabrück
  - RoMed Klinikum Rosenheim, Rosenheim
  - SRH-Klinikum Zentralklinikum Suhl, Suhl
  - Universitätsklinikum Tübingen, Tübingen
- Rijnstate Hospital, Arnhem, Netherlands
- Skane University Hospital, Malmo, Sweden

RESULTS

PARTICIPANT FLOW:
Groups:
- BioMimics 3D Stent: Implantation of BioMimics 3D nitinol stent onto subjects who receive a treatment in accordance with the current approved CE mark indication for use as stated in the IFU.
Period: Overall Study
Arm/Group | BioMimics 3D Stent
Started | 507
30 Days Follow-up | 483
12 Month Follow-up | 418
24 Month Follow-up | 398
Completed | 398
Not Completed | 109
Not completed — Death | 52
Not completed — Lost to Follow-up | 4
Not completed — Withdrawal by Subject | 20
Not completed — Missed Visit | 33

BASELINE CHARACTERISTICS:
Arm/Group | BioMimics 3D Stent
Number analyzed (Participants) | 507
Age, Continuous [Mean (Standard Deviation); unit: Years] | 70.1 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 175
  Male | 332
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 507
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 504
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  Netherlands | 1
  Sweden | 13
  Belgium | 80
  Germany | 413

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Free From Major Adverse Events (MAE)
Description: Primary Safety Endpoint: Number of participants free from a composite of major adverse events (MAE) comprising death, any major amputation performed on the index limb or clinically-driven target lesion revascularization (CDTLR) through 30 days.
Time Frame: 30 days
Population: Participants who came for any follow-up visit (30D, 12M, 24M, 36M) or anyone who experienced a MAE ≤30 days. Twelve (12) participants were ineligible for the primary safety endpoint analysis.
Measure: Count of Participants; unit: Participants
Groups:
- Primary Safety Endpoint: Participants who are free from MAE (death, major amputation on index limb and CDTLR) through 30 days.
Arm/Group | Primary Safety Endpoint
Number analyzed (Participants) | 495
Participants
  30 Days Freedom from MAE | 489
  30 Days Freedom from Death: number analyzed (Participants) | 494
  30 Days Freedom from Death | 492
  30 Days Freedom from Amputation: number analyzed (Participants) | 494
  30 Days Freedom from Amputation | 492
  30 Days Freedom from CDTLR: number analyzed (Participants) | 493
  30 Days Freedom from CDTLR | 491

2. Primary Outcome: Number of Participants Free From Clinically-driven Target Lesion Revascularization (CDTLR)
Description: Primary Effectiveness Endpoint: Number of participants free from clinically-driven target lesion revascularization (CDTLR) through 12 months.
Time Frame: 12 months
Population: Participants who came for a follow-up visit (12M, 24M, 36M) or any participant who experienced CDTLR ≤ 365 days. Sixty-four (64) participants were ineligible for the primary effectiveness endpoint analysis.
Measure: Count of Participants; unit: Participants
Groups:
- Primary Effectiveness Endpoint: Participants free from CDTLR through 12 months.
Arm/Group | Primary Effectiveness Endpoint
Number analyzed (Participants) | 443
Participants | 396

3. Secondary Outcome: Number of Participants With a Final Residual Diameter Stenosis ≤30% at the End of the Index Procedure
Description: Acute Technical Success: Number of participants with a final residual diameter stenosis ≤30% within 72 hours of the index procedure.
Time Frame: Within 72 hours of the index procedure.
Population: One (1) participant did not have a final diameter stenosis recorded at Index, therefore ineligible for acute technical success analysis.
Measure: Count of Participants; unit: Participants
Groups:
- Acute Technical Success: Participants with a final diameter stenosis recorded at Index.
Arm/Group | Acute Technical Success
Number analyzed (Participants) | 506
Participants | 501

4. Secondary Outcome: Number of Participants With Acute Technical Success and Absence of the Adverse Events Listed in the Description
Description: Acute Procedural Success: Number of participants with acute technical success (achievement of a final stenosis ≤30% at the end of the procedure) and absence of the following adverse events: death, stroke, myocardial infarction, acute onset of limb ischemia, index bypass graft or treated segment thrombosis, and/or need for urgent/emergent vascular surgery, within 72 hours of index procedure.
Time Frame: Within 72 hours of index procedure.
Population: All enrolled participants (507) were eligible for acute procedural success analysis.
Measure: Count of Participants; unit: Participants
Groups:
- Acute Procedural Success: Participants who had acute technical success and the absence of the following adverse events: death, stroke, MI, acute onset of limb ischemia, index bypass graft or treated segment thrombosis, and/or need for urgent/emergent vascular surgery, within 72 h of the index procedure.
Arm/Group | Acute Procedural Success
Number analyzed (Participants) | 507
Participants | 494

5. Secondary Outcome: Percent Probability of Individual Components of MAE
Description: A Kaplan-Meier (KM) analysis of individual components of MAE (death, any major amputation performed on the index limb or CDTLR) through 24 months.
Time Frame: 30 days, 12 Months, and 24 Months.
Population: All enrolled participants (507) were eligible for KM analysis of MAE.
Measure: Number; unit: percentage probability
Groups:
- Percent Probability of Individual Components of MAE: Kaplan-Meier analysis of the incidence of death, any major amputation performed on the index limb or CDTLR in the participant population through 24 months.
Arm/Group | Percent Probability of Individual Components of MAE
Number analyzed (Participants) | 507
percentage probability
  KM analysis of Death at 30 Days % | 0.4
  KM analysis of Amputation at 30 Days % | 0.4
  KM analysis of CDTLR at 30 Days % | 0.4
  KM analysis of Death at 12 Months (Day 360) % | 6.1
  KM analysis of Amputation at 12 Months (Day 360) % | 1.5
  KM analysis of CDTLR at 12 Months (Day 360) % | 9.4
  KM analysis of Death at 24 Months (Day 720) % | 10.4
  KM analysis of Amputation at 24 Months (Day 720) % | 1.5
  KM analysis of CDTLR at 24 Months (Day 720) % | 17.2

6. Secondary Outcome: Number of Participants With Adverse Events
Description: Overall rate of all adverse events reported from Day 0 through 24 months. An adverse event (AE) is any untoward medical occurrence, unintended disease or injury, or untoward clinical signs in participants, whether or not related to the investigational device or procedure. For the purpose of this Study all potentially device-related and procedure-related adverse events, major adverse events (death, major amputation on the target limb, clinically-driven target lesion revascularisation), all vascular adverse events in the target limb, and serious adverse events are reported throughout the Study.
Time Frame: 30 day, 12 and 24 months
Population: All enrolled participants (507) were eligible for the rate of AE analysis.
Measure: Count of Participants; unit: Participants
Groups:
- Overall Rate of Adverse Events: Total number of adverse events experienced by the participant population throughout the course of the study.
Arm/Group | Overall Rate of Adverse Events
Number analyzed (Participants) | 507
Participants
  30 Day (≤ 37 days) Participant's Overall Adverse Events | 84
  30 Day (≤ 37 days) Participant's Overall Device Related Adverse Events | 7
  30 Day (≤ 37 days) Participant's Overall Procedure Adverse Events | 36
  30 Day (≤ 37 days) Participant's Overall Serious Adverse Events | 60
  30 Day (≤ 37 days) Participant's Overall Device Related Serious Adverse Events | 6
  30 Day (≤ 37 days) Participant's Overall Procedure Related Serious Adverse Events | 21
  12 Month (≤ 395 days) Participant's Overall Adverse Events | 255
  12 Month (≤ 395 days) Participant's Overall Device Related Adverse Events | 67
  12 Month (≤ 395 days) Participant's Overall Procedure Related Adverse Events | 68
  12 Month (≤ 395 days) Participant's Overall Serious Adverse Events | 219
  12 Month (≤ 395 days) Participant's Overall Device Related Serious Adverse Events | 59
  12 Month (≤ 395 days) Participant's Overall Procedure Related Serious Adverse Events | 44
  24 Month (≤ 790 days) Participant's Overall Adverse Events | 318
  24 Month (≤ 790 days) Participant's Overall Device Related Adverse Events | 93
  24 Month (≤ 790 days) Participant's Overall Procedure Related Adverse Events | 74
  24 Month (≤ 790 days) Participant's Overall Serious Adverse Events | 282
  24 Month (≤ 790 days) Participant's Overall Device Related Serious Adverse Events | 79
  24 Month (≤ 790 days) Participant's Overall Procedure Related Serious Adverse Events | 50

7. Secondary Outcome: Stent Patency Rate
Description: Per Protocol, patency is defined as the composite of freedom from more than 50% restenosis within the stented segment as observed by Duplex Ultrasound or Angiography within the visit window and freedom from clinically-driven target lesion revascularisation prior to the indicated time point. Stent patency rate assessed by duplex ultrasound (DUS), as available, determined at Months 12 and 24. This will be assessed using values of peak systolic velocity ratio (PSVR) >2.0, >2.4; >2.5; and >3.5. PSVR values of >2.0, >2.4, >2.5 and >3.5 were selected to compare outcomes from similar studies. There are no official definitions or guidelines on these values and which are most accurate for detection of >50% stenosis, so all have been used in the analyses to compare results from other studies. PSVR of >2.4, was looked at further as there are some studies that state this is the most established threshold for the detection of >50% stenosis (Schlager, et al. 2007).
Time Frame: 12 and 24 months.
Population: Number of participants who had patency assessed at month 12 was 443. Number of participants who had patency assessed at month 24 was 409.
Measure: Count of Participants; unit: Participants
Groups:
- Stent Patency: Participants who have a duplex ultrasound at month 12 or 24 will have stent patency assessed using PSVR values >2.0, >2.4, >2.5, and >3.5, each to indicate loss of patency on duplex ultrasound.
Arm/Group | Stent Patency
Number analyzed (Participants) | 443
Participants
  Patency at 12 Months PSVR >2.0 | 370
  Patency at 12 Months PSVR >2.4 | 381
  Patency at 12 Months PSVR >2.5 | 381
  Patency at 12 Months PSVR >3.5 | 388
  Patency at 24 Months PSVR >2.0: number analyzed (Participants) | 409
  Patency at 24 Months PSVR >2.0 | 318
  Patency at 24 Months PSVR >2.4: number analyzed (Participants) | 409
  Patency at 24 Months PSVR >2.4 | 324
  Patency at 24 Months PSVR >2.5: number analyzed (Participants) | 409
  Patency at 24 Months PSVR >2.5 | 324
  Patency at 24 Months PSVR >3.5: number analyzed (Participants) | 409
  Patency at 24 Months PSVR >3.5 | 324

8. Secondary Outcome: Comparison of Rutherford Clinical Category
Description: Clinical Outcome: Comparison of Rutherford Clinical Category (RCC) measured at Baseline, Day 30, Months 12 and 24. Rutherford Clinical Category is a clinical scale identifying three grades of claudication (RCC 1-3) and three grades of critical limb ischemia (RCC 4-6) ranging from rest pain alone to minor and major tissue loss. Category and clinical description: 0 - Asymptomatic, 1 - Mild claudication 2 - Moderate claudication, 3 - Severe claudication, 4 - Ischemic rest pain, 5 - Minor tissue loss, 6 - Ulceration or gangrene.
Time Frame: Baseline, Day 30, 12 months and 24 months
Population: RCC is collected serially over time and is presented at each time point. The measure from each time point is compared to the baseline measure. Three (3) participants did not have a baseline RCC assessed.
Measure: Count of Participants; unit: Participants
Groups:
- Rutherford Clinical Category: Comparing participants Rutherford Clinical Category (RCC) from Baseline to day 30, months 12 and 24.
  Claudication - RCC 1, 2, 3. Critical Limb Ischemia - RCC 4, 5, 6.
Arm/Group | Rutherford Clinical Category
Number analyzed (Participants) | 504
Participants
  Baseline RCC 0 | 2
  Baseline RCC 1 | 6
  Baseline RCC 2 | 86
  Baseline RCC 3 | 289
  Baseline RCC 4 | 38
  Baseline RCC 5 | 72
  Baseline RCC 6 | 11
  30 Days RCC 0: number analyzed (Participants) | 423
  30 Days RCC 0 | 172
  30 Days RCC 1: number analyzed (Participants) | 423
  30 Days RCC 1 | 121
  30 Days RCC 2: number analyzed (Participants) | 423
  30 Days RCC 2 | 62
  30 Days RCC 3: number analyzed (Participants) | 423
  30 Days RCC 3 | 30
  30 Days RCC 4: number analyzed (Participants) | 423
  30 Days RCC 4 | 7
  30 Days RCC 5: number analyzed (Participants) | 423
  30 Days RCC 5 | 30
  30 Days RCC 6: number analyzed (Participants) | 423
  30 Days RCC 6 | 1
  12 Months RCC 0: number analyzed (Participants) | 375
  12 Months RCC 0 | 151
  12 Months RCC 1: number analyzed (Participants) | 375
  12 Months RCC 1 | 121
  12 Months RCC 2: number analyzed (Participants) | 375
  12 Months RCC 2 | 60
  12 Months RCC 3: number analyzed (Participants) | 375
  12 Months RCC 3 | 36
  12 Months RCC 4: number analyzed (Participants) | 375
  12 Months RCC 4 | 4
  12 Months RCC 5: number analyzed (Participants) | 375
  12 Months RCC 5 | 2
  12 Months RCC 6: number analyzed (Participants) | 375
  12 Months RCC 6 | 1
  24 Months RCC 0: number analyzed (Participants) | 345
  24 Months RCC 0 | 130
  24 Months RCC 1: number analyzed (Participants) | 345
  24 Months RCC 1 | 123
  24 Months RCC 2: number analyzed (Participants) | 345
  24 Months RCC 2 | 48
  24 Months RCC 3: number analyzed (Participants) | 345
  24 Months RCC 3 | 38
  24 Months RCC 4: number analyzed (Participants) | 345
  24 Months RCC 4 | 3
  24 Months RCC 5: number analyzed (Participants) | 345
  24 Months RCC 5 | 2
  24 Months RCC 6: number analyzed (Participants) | 345
  24 Months RCC 6 | 1

9. Secondary Outcome: Comparison of Ankle Brachial Index (ABI) Measurement
Description: Functional outcome: Mean and standard deviation of the Ankle Brachial Index at each follow-up visit is reported.
  The change of Ankle Brachial Index at 30 days, 12 and 24 months compared to Baseline is presented for the total number of patients where data were recorded, and the mean and standard deviation of the change.
  ABI is the ratio of blood pressure measured at the ankle to blood pressure measured at the arms. It is used to predict the severity of peripheral arterial disease. An ABI of >0.9-1.2 is considered normal, ≤ 0.9 indicates mild to moderate peripheral arterial disease, < 0.4 indicates severe peripheral arterial disease (ischemic pain and ulceration).
Time Frame: Baseline, Day 30, 12-month and 24-month.
Population: Four-hundred and seventeen (417) participants had their ABI measured at Baseline. Three-hundred and eighty-three (383) participants at Day 30. Three hundred and fifty-nine (359) participants at Month 12. Three-hundred and four participants at Month 24.
Measure: Mean (Standard Deviation); unit: ABI
Groups:
- Ankle Brachial Index Measurement: Comparison of the ABI measurement from Baseline, Day 30, Months 12 and 24.
Arm/Group | Ankle Brachial Index Measurement
Number analyzed (Participants) | 417
ABI
  Baseline ABI | 0.6 (0.30)
  30 Days ABI: number analyzed (Participants) | 383
  30 Days ABI | 1.0 (0.2)
  12 Months ABI: number analyzed (Participants) | 359
  12 Months ABI | 0.9 (0.2)
  24 Months ABI: number analyzed (Participants) | 304
  24 Months ABI | 0.9 (0.2)
  30 Days Change from Baseline ABI: number analyzed (Participants) | 348
  30 Days Change from Baseline ABI | 0.4 (0.3)
  12 Months Change from Baseline ABI: number analyzed (Participants) | 319
  12 Months Change from Baseline ABI | 0.3 (0.3)
  24 Months Change from Baseline ABI: number analyzed (Participants) | 270
  24 Months Change from Baseline ABI | 0.3 (0.3)

10. Secondary Outcome: Number of Participants With Reported Stent Fracture
Description: Site reported number of participants with stent fracture through 24 months. Stent fracture is defined as clear interruption of stent strut observed in a minimum of two projections, determined by examination of X-ray images.
  Stent Strut Fracture Types: Type 0: No strut fractures. Type I: Single strut fracture only. Type II: Multiple single strut fractures that can occur at different sites. Type III: Multiple strut fractures resulting in complete transection of the stent, without displacement of the stent segments. Type IV: Multiple strut fractures resulting in displacement of segments of the stent. Type V: Spiral strut fracture.
Time Frame: 30 day, 12 and 24 Months.
Population: Four-hundred and eighty-three (483) participants were eligible for this analysis at Day 30; 418 at Month 12; 398 at Month 24. Five (5) participants had X-ray images obtained at Day 30; 5 participants had X-ray images obtained at Month 12; 3 participants had X-ray images obtained at Month 24. In an observational registry x-rays are only conducted if there are clinical symptoms that hint towards a fracture. In the absence of symptoms it is concluded that the subject did not suffer a stent fracture
Measure: Count of Participants; unit: Participants
Groups:
- Number of Participants With Reported Stent Fracture: Site reported number of participants who have a reported stent fracture through the 24-month timepoint.
Arm/Group | Number of Participants With Reported Stent Fracture
Number analyzed (Participants) | 483
Participants
  Stent Fracture at 30 Days | 0
  Stent Fracture at 12 Months: number analyzed (Participants) | 418
  Stent Fracture at 12 Months | 0
  Stent Fracture at 24-Months: number analyzed (Participants) | 398
  Stent Fracture at 24-Months | 3
  Stent Fracture Category Type 0 at 24 Months: number analyzed (Participants) | 398
  Stent Fracture Category Type 0 at 24 Months | 0
  Stent Fracture Category Type I at 24 Months: number analyzed (Participants) | 398
  Stent Fracture Category Type I at 24 Months | 0
  Stent Fracture Category Type II at 24 Months: number analyzed (Participants) | 398
  Stent Fracture Category Type II at 24 Months | 3
  Stent Fracture Category Type III at 24 Months: number analyzed (Participants) | 398
  Stent Fracture Category Type III at 24 Months | 0
  Stent Fracture Category Type IV at 24 Months: number analyzed (Participants) | 398
  Stent Fracture Category Type IV at 24 Months | 0
  Stent Fracture Category Type V at 24 Months: number analyzed (Participants) | 398
  Stent Fracture Category Type V at 24 Months | 0

ADVERSE EVENTS:
Time Frame: 24 months
Description: AE reported by sites & required to be reported to the Sponsor within 24 hrs of knowledge of the AE or by the end of the next working day as defined in the Protocol are:
  * All potentially device &/or procedure-related AE
  * All major adverse events (MAE)
  * All vascular AE in the target limb
  * SAE "Other events" describe AE that do not have an AE code that is prepopulated on the database. These AE were monitored and assessed using the same processes that AE with the prepopulated AE code were.
Groups:
- Implantation of BioMimics 3D Nitinol Stent: Implantation of BioMimics 3D nitinol stent using the BioMimics 3D Stent System
Arm/Group | Implantation of BioMimics 3D Nitinol Stent
All-Cause Mortality (participants affected / at risk) | 52/507
Serious Adverse Events (participants affected / at risk) | 282/507
Other Adverse Events (participants affected / at risk) | 19/507
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Implantation of BioMimics 3D Nitinol Stent (N=507)
Allergic reaction (Immune system disorders) | 1 (1)
Amputation unplanned (Vascular disorders) | 11 (13)
Aneurysm (Vascular disorders) | 5 (6)
Arterial stenosis (non-target, de novo) (Vascular disorders) | 43 (45)
Embolization, distal (Vascular disorders) | 3 (3)
Necrosis (Vascular disorders) | 1 (1)
Occlusion, early (Vascular disorders) | 1 (1) — (less than 30 days treated vessel)
Occlusion, other (Vascular disorders) | 54 (66)
Pseudoaneurysm (target vessel) (Vascular disorders) | 1 (1)
Pseudoaneurysm (access site) (Vascular disorders) | 5 (5)
Restenosis of treated segment, target lesion (Vascular disorders) | 66 (80)
Restenosis of treated vessel, target vessel (Vascular disorders) | 12 (13)
Restenosis, non-target vessel or region (Vascular disorders) | 20 (22)
Thrombosis (treated segment) (Vascular disorders) | 5 (7)
Anemia (Blood and lymphatic system disorders) | 5 (5)
Bleeding from anticoagulant or antiplatelet meds (Blood and lymphatic system disorders) | 1 (1)
Angina (Cardiac disorders) | 6 (11)
Atrial fibrillation (Cardiac disorders) | 6 (6)
Cardiac arrhythmia (excl. AFib) (Cardiac disorders) | 3 (3)
Cardiopulmonary arrest (Cardiac disorders) | 1 (1)
Congestive heart failure (Cardiac disorders) | 10 (10)
Hypertension (Cardiac disorders) | 2 (2)
Myocardial infarction (Cardiac disorders) | 8 (8)
Myocardial ischemia (Cardiac disorders) | 5 (5)
Other ischemia (Cardiac disorders) | 3 (3)
Arterial occlusion/thrombus at puncture site (Injury, poisoning and procedural complications) | 3 (3)
Groin hematoma greater or equal to 5cm, with or without surgical repair (Injury, poisoning and procedural complications) | 1 (1)
Other access site complication requiring surgery or transfusion (Injury, poisoning and procedural complications) | 1 (1)
Pain or discomfort at access site (greater than 24h after procedure) (Injury, poisoning and procedural complications) | 1 (1)
Fever (higher than 38.3ºC/101ºF) (General disorders) | 2 (2)
Gastro-intestinal bleeding (Gastrointestinal disorders) | 8 (9)
Infected peripheral wound (Infections and infestations) | 5 (5)
Infection, access site (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 7 (7)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 9 (10)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 7 (8)
Renal failure/renal insufficiency (Renal and urinary disorders) | 4 (4)
Stroke (Nervous system disorders) | 6 (6)
Other event (Investigations) | 112 (159) — Other events
Limb Ischemia (Vascular disorders) | 1 (1)
Bacteremia or septicemia (Infections and infestations) | 1 (1)
Amputation (planned) (Vascular disorders) | 7 (9)
Pseudoaneurysm, other (Vascular disorders) | 4 (4)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Implantation of BioMimics 3D Nitinol Stent (N=507)
Occlusion, other (Vascular disorders) | 8 (8)
Restenosis of treated segment (target lesion) (Vascular disorders) | 11 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-03): https://cdn.clinicaltrials.gov/large-docs/24/NCT02900924/Prot_SAP_000.pdf